CLINICAL TRIAL: NCT05928325
Title: Implementation of a Geriatric Care Survivorship Intervention in Older Adults Who Have Completed Curative Intent Therapy for Early-Stage Breast Cancer
Brief Title: Geriatric Care Survivorship Intervention for Improving the Overall Health of Older Adults With Stage I-III Breast Cancer Who Have Completed Curative Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-1125; NCI-2022-00935 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1125 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8
MeSH Terms: interventions — Geriatric Assessment; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (GA-guided intervention) (Experimental): Patients complete geriatric assessments at baseline, 6 months, and 12 months later. Based on the assessments, patients may receive further intervention at survivorship visit. Patients also receive survivorship care educational materials and wear a wearable activity tracking device for 1 year on study.
  Interventions: Other: Comprehensive Geriatric Assessment; Behavioral: Health Education; Other: Medical Device Usage and Evaluation; Other: Supportive Care

INTERVENTIONS:
Other: Comprehensive Geriatric Assessment — Complete geriatric assessments
Behavioral: Health Education — Receive survivorship care education
Other: Medical Device Usage and Evaluation — Wear activity tracking device
Other: Supportive Care — Receive geriatric assessment-guided interventions
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive

SUMMARY:
This trial studies the effect of a geriatric care survivorship intervention in improving the overall health of older adults who have completed curative treatment for stage I-III breast cancer. Geriatric assessment is the complete examination of an elderly individual, which includes a full valuation of the physical and mental conditions, as well as a check of emotional state. Geriatric assessment and survivorship visits after treatment may reduce health burdens and improve the well-being and quality of life of elderly patients with breast cancer. Researchers hope to improve the overall health of older adults who have undergone curative treatment for stage I-III breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the feasibility of implementing the geriatric care survivorship intervention in older adults who have completed curative-intent chemotherapy.

SECONDARY OBJECTIVES:

I. Assess the impact of a Geriatric Assessment (GA)-guided intervention on patient-reported quality-of-life/physical function (assessed by the Functional Assessment of Cancer Therapy-Breast [FACT-B]), geriatric assessment measures (assessed by GA) and objective physical function (assessed by the Short Physical Performance Battery [SPPB]) in older survivors from baseline to 6- and 12-months +/- 4-weeks post-chemotherapy.

II. Determine the impact of intervention on patient reported cognitive function (FACT-Cog) and objective cognitive function (Mini-Cog) from baseline to 6- and 12-months +/- 4-weeks post-chemotherapy.

III. Estimate the effect of the intervention on completion of referral appointments and contacts with primary care providers.

IV. Estimate the effect of the intervention on emergent healthcare utilization (emergency room [ER] visits and hospitalizations) at 6- and 12-months +/- 4 weeks post-chemotherapy.

V. Determine the impact of the intervention on both patient and caregiver satisfaction with care ("Health Care Climate Questionnaire") from baseline to 6- and 12-months +/- 4-weeks post-chemotherapy.

VI. Determine the impact of intervention on caregiver distress ("Burden Scale for Family Caregivers") and satisfaction with care ("Health Care Climate Questionnaire") from baseline to 6- and 12-months +/- 4-weeks post-chemotherapy.

OUTLINE:

Patients complete geriatric assessments at baseline, 6 months, and 12 months later. Based on the assessments, patients may receive further intervention at survivorship visit. Patients also receive survivorship care educational materials and wear a wearable activity tracking device for 1 year on study.

ELIGIBILITY:
Inclusion Criteria:

* >= 65-years-old
* Histologically confirmed Stage I, II or III breast cancer (if the patient has had more than one breast cancer, the most recent diagnosis)
* Within 8 (+/- 14 days) weeks of completing a chemotherapy regimen for breast cancer either as standard-of-care or on a study (can be receiving concomitant radiation, HER-2 targeted agents and/or endocrine therapy)
* English or Spanish speaking
* Able to provide written, informed consent
* Willing and able to meet all study requirement
* CAREGIVER ELIGIBILITY: >= 18-years-old
* CAREGIVER ELIGIBILITY: Ability to complete required study procedures

Exclusion Criteria:

* The presence of significant medical conditions that in the physician's (either the patient's primary oncologist of the study principal investigator) judgement preclude participation in the exercise intervention

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy-Breast (FACT-B) questionnaires | through study completion; an average of 1 year.
  The FACT-G is a 27-item instrument that uses a 5-point Likert-type scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much).

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Karuturi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://mdanderson.org